CLINICAL TRIAL: NCT03405220
Title: Testing a Self-affirmation Intervention for Use in a Mobile Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kent State University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jennifer Taber, Assistant Professor, Kent State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-544
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Smoking; Smoking Cessation; Smoking, Tobacco
Keywords: smoking; self-affirmation; mobile application; cessation
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Study 1 will use a 2 (self-affirmation: self-affirmation, control) X 3 (Mode of example: none, write, imagine) experimental design. In the self-affirmation condition, participants will complete the self-affirmation kindness quiz (10 questions) and in the control condition they will complete a personal opinion survey (10 questions). Depending on the mode of example condition, participants will not be asked to provide examples, asked to write examples for each of the 10 questions, or asked to imagine examples for each of the 10 questions.
  Based on examination of data from Study 1 (i.e., which items receive more "yes" responses and for which items examples are provided), in Study 2 we will test whether using fewer self-affirmation items influences dependent variables. Study 2 will use a 3 (Number of questions: 10, 5, 3) X 3 (Mode of example: none, write, imagine) experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Self-affirm, No examples, Study 1 (Experimental): Behavioral: Self affirmation, 10 items, no examples
  Interventions: Behavioral: Self affirmation, 10 items, no examples
- Self-affirm, Write examples, Study 1 (Active Comparator): Behavioral: Self affirmation, 10 items, written examples
  Interventions: Behavioral: Self affirmation, 10 items, written examples
- Self-affirm, Imagine examples, Study 1 (Experimental): Behavioral: Self affirmation, 10 items, imagined examples
  Interventions: Behavioral: Self affirmation, 10 items, imagined examples
- Opinion survey, No examples, Study 1 (No Intervention): No intervention: control. Participants will complete the 10 item personal opinion survey and will not be asked to provide examples for any items they respond "yes" to.
- Opinion survey, Write examples, Study 1 (No Intervention): No intervention: control. Participants will complete the 10 item personal opinion survey and will be asked to provide written examples for each item they respond "yes" to.
- Opinion survey, Imagine examples, Study1 (No Intervention): No intervention: control. Participants will complete the 10 item personal opinion survey and will be asked to imagine examples for each item they respond "yes" to.
- Self-affirm, 10-item, No ex, Study 2 (Experimental): Behavioral: Self affirmation, 10 items, no examples
  Interventions: Behavioral: Self affirmation, 10 items, no examples
- Self-affirm, 5-item, No ex, Study 2 (Experimental): Behavioral: Self affirmation, 5 items, no examples
  Interventions: Behavioral: Self affirmation, 5 items, no examples
- Self-affirm, 3-item, No ex, Study 2 (Experimental): Behavioral: Self affirmation, 3 items, no examples
  Interventions: Behavioral: Self affirmation, 3 items, no examples
- Self-affirm, 10-item, Write ex, Study 2 (Active Comparator): Behavioral: Self affirmation, 10 items, written examples
  Interventions: Behavioral: Self affirmation, 10 items, written examples
- Self-affirm, 5-item, Write ex, Study 2 (Experimental): Behavioral: Self affirmation, 5 items, written examples
  Interventions: Behavioral: Self affirmation, 5 items, written examples
- Self-affirm, 3-item, Write ex, Study 2 (Experimental): Behavioral: Self affirmation, 3 items, written examples
  Interventions: Behavioral: Self affirmation, 3 items, written examples
- Self-affirm, 10-item, Imagine ex, Study2 (Experimental): Behavioral: Self affirmation, 10 items, imagined examples
  Interventions: Behavioral: Self affirmation, 10 items, imagined examples
- Self-affirm, 5-item, Imagine ex, Study 2 (Experimental): Behavioral: Self affirmation, 5 items, imagined examples
  Interventions: Behavioral: Self affirmation, 5 items, imagined examples
- Self-affirm, 3-item, Imagine ex, Study 2 (Experimental): Behavioral: Self affirmation, 3 items, imagined examples
  Interventions: Behavioral: Self affirmation, 3 items, imagined examples

INTERVENTIONS:
Behavioral: Self affirmation, 10 items, written examples — Participants will complete the 10 item self-affirmation kindness quiz and will be asked to provide written examples for each item they respond "yes" to.
  Arms: Self-affirm, 10-item, Write ex, Study 2; Self-affirm, Write examples, Study 1
Behavioral: Self affirmation, 10 items, no examples — Participants will complete the 10 item self-affirmation kindness quiz and will not be asked to provide examples for any items they respond "yes" to.
  Arms: Self-affirm, 10-item, No ex, Study 2; Self-affirm, No examples, Study 1
Behavioral: Self affirmation, 10 items, imagined examples — Participants will complete the 10 item self-affirmation kindness quiz and will be asked to imagine examples for each item they respond "yes" to.
  Arms: Self-affirm, 10-item, Imagine ex, Study2; Self-affirm, Imagine examples, Study 1
Behavioral: Self affirmation, 5 items, written examples — Participants will complete a 5 item self-affirmation kindness quiz and will be asked to provide written examples for each item they respond "yes" to.
  Arms: Self-affirm, 5-item, Write ex, Study 2
Behavioral: Self affirmation, 5 items, no examples — Participants will complete a 5 item self-affirmation kindness quiz and will not be asked to provide examples for any items they respond "yes" to.
  Arms: Self-affirm, 5-item, No ex, Study 2
Behavioral: Self affirmation, 5 items, imagined examples — Participants will complete a 5 item self-affirmation kindness quiz and will be asked to imagine examples for each item they respond "yes" to.
  Arms: Self-affirm, 5-item, Imagine ex, Study 2
Behavioral: Self affirmation, 3 items, written examples — Participants will complete a 3 item self-affirmation kindness quiz and will be asked to provide written examples for each item they respond "yes" to.
  Arms: Self-affirm, 3-item, Write ex, Study 2
Behavioral: Self affirmation, 3 items, no examples — Participants will complete a 3 item self-affirmation kindness quiz and will not be asked to provide examples for any items they respond "yes" to.
  Arms: Self-affirm, 3-item, No ex, Study 2
Behavioral: Self affirmation, 3 items, imagined examples — Participants will complete a 3 item self-affirmation kindness quiz and will be asked to imagine examples for each item they respond "yes" to.
  Arms: Self-affirm, 3-item, Imagine ex, Study 2

SUMMARY:
The aim of these studies is to adapt the self-affirmation kindness questionnaire for use in a mobile application. Two studies will be conducted to test hypotheses that simplifying and shortening the original questionnaire in systematic ways will result in comparable effectiveness (compared to the original version) in promoting reduced defensive avoidance, less reactance, greater yielding, and higher intentions to quit smoking among a sample of smokers.

DETAILED DESCRIPTION:
Research has shown that self-affirmation interventions, in which people are instructed to focus on their strengths and values, can offset self-threats and promote healthier behaviors, such as smoking cessation. A commonly used self-affirmation intervention is known as the "kindness quiz." The original kindness questionnaire (Reed & Aspinwall, 1998) consists of 10 yes/no questions, and participants are asked to think about and write down an example of each. For example, one item is "Have you ever been considerate of another person's feelings? ____ YES ____NO; IF YES, WRITE ABOUT A SPECIFIC EXAMPLE." The items were written so that all participants should be able to say "yes" in response to each question, which will affirm a positive view of themselves.

The purpose of these studies are to test shorter and simpler versions of this kindness questionnaire so that it can be implemented on mobile phones. In Study 1, we will test whether written examples are necessary for the effectiveness of the self-affirmation intervention (compared to no examples or imagined examples) compared to a control. In Study 2, we will again test whether written examples are necessary, as well as whether shorter questionnaires (i.e., 5 items or 3 items) are as effective as the original 10 item questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Currently live in the US
* 21-65 years (several states have 21 as minimum legal age to smoke)
* self-identified every day or some day smoker
* no prior diagnosis of lung cancer, chronic obstructive pulmonary disease, or emphysema (the most common and well-known smoking-related diseases

Exclusion Criteria:

* Not currently living in the US
* Less than 21 years of age or older than 65
* Nonsmoker
* Prior diagnosis of lung cancer, chronic obstructive pulmonary disease, or emphysema (the most common and well-known smoking-related diseases

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Defensive Avoidance | immediately post-intervention
  Indicator of defensive information processing, 3 items (Witte)
Reactance | immediately post-intervention
  Indicator of defensive information processing, 27 items (Hall et al., 2016)
Yielding | immediately post-intervention
  Indicator of defensive information processing, 7 items (Brennan et al., 2011, 2014)
Intentions to quit smoking in the next 3 months | immediately post-intervention
  Intentions to quit smoking, 3 items

SECONDARY OUTCOMES:
Cognitive perceived likelihood of developing smoking related disease | immediately post-intervention
  3 items
Perceived severity | immediately post-intervention
  3 items
Response efficacy of quitting smoking | immediately post-intervention
  3 items
Self-efficacy to quit smoking | immediately post-intervention
  3 items
Affective perceived likelihood | immediately post-intervention
  3 items
Anticipated regret | immediately post-intervention
  3 items
Worry | immediately post-intervention
  3 items

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Taber, PhD, Principal Investigator — Kent State University
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be made available to other researchers upon request following publication of the results of the study. Alternatively, data may be posted on a site such as Open Science Framework and made publicly available.

REFERENCES:
- [Background] Reed, M. B., & Aspinwall, L. G. (1998). Self-affirmation reduces biased processing of health-risk information. Motivation and Emotion, 22(2), 99-132.

DOCUMENTS (1):
  • Informed Consent Form (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03405220/ICF_000.pdf